CLINICAL TRIAL: NCT04595825
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Clinical Trial Evaluating the Safety and Efficacy of CM-101 in Subjects With Primary Sclerosing Cholangitis (The SPRING Study)
Brief Title: CM-101 in PSC Patients -The SPRING Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-PSC-101
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Anti-fibrotic
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anti-human CCL24 monoclonal antibody (CM-101) (Experimental): Anti-human CCL24 monoclonal antibody CM-101 Intravenous Infusion over 60 minutes (±5 minutes)
  Interventions: Biological: Anti-human CCL24 monoclonal antibody (CM-101)
- Placebo (Placebo Comparator): Placebo - intravenous infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Anti-human CCL24 monoclonal antibody (CM-101) — Anti-human CCL24 monoclonal antibody (CM-101) 100 mg Intravenous Infusion over 60 minutes (±5 minutes)
  Arms: Anti-human CCL24 monoclonal antibody (CM-101)
Other: Placebo — Placebo - intravenous infusion
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety, tolerability and activity of the anti-human CCL24 monoclonal antibody CM-101 in adult subjects with Primary Sclerosing Cholangitis (PSC). At least 68 subjects at approximately 50 sites will be randomized to receive either CM-101 at doses of 10 mg/kg or 20 mg/kg or matching placebo.

DETAILED DESCRIPTION:
This study will consist of a screening period, double-blind (DB) treatment period, open-label (OL) treatment period, and safety follow-up period. During the DB treatment period, subjects will receive 5 total dose administrations of study drug (investigational product - IP or placebo) once every 3 weeks (Q3W) for a coverage of 15 weeks. After completing the DB treatment period, subjects may elect to enroll in an OL treatment period. In the OL treatment period, subjects will receive a dose of IP Q3W for 11 administrations for a coverage of 33 weeks, resulting in a combined total coverage of up to 48 weeks.

Subjects who do not elect to continue treatment in the OL dosing period will undergo an End of Treatment (EOT)-DB visit at Week 15 (Day 105), a Safety Follow-up Call at Week 21 (Day 147), and an End of Study (EOS) visit at Week 27. Eligible subjects who continue treatment in the OL treatment period will receive CM-101 at either a 10 mg/kg or 20 mg/kg dose commencing at Week 15 (OL Treatment 1), and the subjects will undergo an EOT-OL visit at Week 48 (Day 336), a Safety Follow-up Call at Week 54 (Day 378), and an EOS visit at Week 60 (Day 420).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of large duct PSC of more than 24 weeks' duration
* Subjects that have no significant clinical concern for cholangiocarcinoma based on clinical, laboratory or imaging findings
* Subjects with serum Alkaline phosphatase (ALP) greater than 1.5 × Upper limit of normal (ULN) in Screening blood tests.
* Subjects receiving Ursodeoxycholic acid (UDCA) must receive a stable dose for ≥12 weeks prior to Screening
* Subjects with concomitant inflammatory bowel disease (IBD) is allowed but not required, and must meet the following stability criteria.

Subjects with ulcerative colitis: Must be either in remission or have mild disease. Must have recent colonoscopy with biopsy confirming no dysplasia or colorectal cancer or history of colectomy.

* Subjects with Crohn's Disease must be in remission as defined by a Crohn's Disease Activity Index (CDAI) < 150.
* Subjects receiving concomitant medication for IBD, dose must be stable ≥12 weeks prior to screening and dose should remain stable during DB portion of the study

  * Subjects receiving concomitant medication for their PSC must be on stable therapy ≥12 weeks prior to randomization and plan to remain on that stable dose during the DB portion of the study
  * Female subjects of childbearing potential, must have a negative serum pregnancy test prior to starting study treatment and must have agree to highly effective method of contraception from the Screening Visit throughout the study period including 18 weeks post last dose
  * Male subjects, if not vasectomized, must agree to use barrier contraception from screening through to study completion and for 90 days from the last dose of study drug

Exclusion Criteria:

* Subjects with presence of documented secondary sclerosing cholangitis on prior clinical investigations
* Subjects with presence of competing etiology of liver disease.
* Subjects with possible overlap syndrome with autoimmune hepatitis are excluded if the Investigator considers autoimmune hepatitis as the predominant liver injury
* Subjects with small duct PSC in the absence of large duct disease
* Subjects with percutaneous biliary drain or bile duct stent or subjects who had required biliary drainage within 12 weeks of Screening
* Subjects that have undergone prior biliary surgery other than those who at the time of screening are more than 6 weeks after cholecystectomy without surgical complications
* Subjects with evidence of liver cirrhosis, as determined by local transient elastography values of ≥ 14.4 kPa obtained during the Screening period. In case of a fibrosis staging discrepancy between a recent (≤ 12 months) liver biopsy staging and the transient elastography results, eligibility will be based on the liver biopsy staging.
* History of cirrhosis and/or hepatic impairment (Child-Pugh classes A, B and C), and/or hepatic decompensation including ascites, encephalopathy, or variceal bleeding
* Subjects who have undergone or are planned for liver transplantation or with current model of end stage liver disease
* Subjects with Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) values > 5 × ULN as determined at Screening
* Subjects who show 'clinically significant' lab changes at Screening
* Subjects with serum total bilirubin values > 3 × ULN at Screening
* Subjects with known Gilbert's syndrome or a history of elevations in unconjugated (indirect) bilirubin >ULN
* Subjects with international normalized ratio (INR) >1.5 which does not correct on vitamin K replacement, in the absence of anticoagulants
* Subjects with serum creatinine > 1.4 mg/dL (123 μmol/L) and/or a platelet count < 100 × 109 /L
* Subjects with history of cholangiocarcinoma or a high clinical suspicion for cholangiocarcinoma
* Subjects with elevated cancer antigen 19-9 (Ca 19-9) value (> 129 U/mL) within 12 months prior to Screening unless Ca 19-9 levels have been stable and clinical evaluation and repeated Magnetic resonance imaging (MRI) within the same time period has not provided evidence of cholangiocarcinoma
* Subjects with a prior biliary stricture necessitating intervention should be stable for ≥ 24 weeks prior to randomization without intervention, or episode of cholangitis, and should show a low level of clinical suspicion of cholangiocarcinoma
* Subjects with current known portal hypertension with complications, including known gastric or large esophageal varices, poorly controlled or diuretic resistant ascites, history of variceal bleeds, or related therapeutic or prophylactic interventions
* Subjects with active malignancy (diagnosed and/or treated within 3 years of randomization), other than:

  * adequately treated non-metastatic basal cell skin cancer
  * squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to randomization
  * history of cervical carcinoma in situ that has been adequately treated and that has not recurred.
* Subjects with a 'clinically significant' (as judged by the Investigator) unexplained weight loss during the 24 weeks prior to randomization
* Subjects showing deleterious effects of alcohol abuse or that consume excessive amounts of alcohol
* Subjects with known or suspected acute cholangitis in the 90 days prior to randomization, including cholangitis treated with antibiotics within the 90 days
* Subjects experiencing flare in colitis activity within 90 days of randomization requiring intensification of therapy beyond baseline maintenance treatment or use of oral prednisone > 10 mg/day (or equivalent), start or dose change of biologics ≤ 12 weeks before screening and or hospitalization for colitis within 90 days of randomization
* Subjects treated with or who are expected to begin treatment with fenofibrate or other fibrates or subjects who had a change in dose within 24 weeks of Screening, or subjects who are not planned to remain on a stable dose throughout the DB portion of the study
* Subjects that use any prohibited medication
* Subjects who have a known history of hypersensitivity reaction to CHO-derived antibodies, CM-101, or any of the formulation excipients
* Subjects with known chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or that have positive hepatitis B surface antigen (HBSAg) at Screening
* Subjects with evidence of an active infection during the Screening period
* Subjects with any identified congenital or acquired immune-deficiency
* Subjects who have gone through major surgical procedure within 60 days of randomization or have had prior organ transplantation
* Subjects who have received a live/attenuated vaccine within 30 days of study randomization
* Female subjects who are pregnant or breast- feeding
* Subjects that have participated in an investigational trial of a drug or device either within 60 days of randomization; or where the study drug half-life is greater than 12 days, at least 5 half-lives need to have passed from the last dose of investigational drug prior to randomization
* Subjects with any other conditions, clinically significant disorders, or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing and study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety-related endpoints - number of participants with treatment-emergent adverse events (TEAEs) | 15 week double-blind (DB) treatment period
  Frequency and severity of treatment-emergent adverse events (TEAEs), including vital sign changes, changes in clinical safety laboratories and evaluation of infusion site reactions.

SECONDARY OUTCOMES:
Safety-related endpoints - number of participants with abnormal vital sign changes | 48 week double-blind (DB) and open-label (OL) treatment periods
  Frequency and severity of treatment-emergent adverse events (TEAEs), including abnormal vital sign changes.
Safety-related endpoints - number of participants with abnormal changes in clinical safety laboratory test results | 48 week double-blind (DB) and open-label (OL) treatment periods
  Frequency and severity of treatment-emergent adverse events (TEAEs), including changes in clinical safety laboratories.
Safety-related endpoints - number of participants with infusion site reactions | 48 week double-blind (DB) and open-label (OL) treatment periods
  Frequency and severity of treatment-emergent adverse events (TEAEs), including evaluation of infusion site reactions.
Alkaline phosphate (ALP) levels | Change from baseline through Week 15
  Serum ALP levels by treatment cohort
Enhanced Liver Fibrosis (ELF) score value | Change from baseline through Week 15
  ECM marker set consisting of tissue inhibitor of metalloproteinases 1 (TIMP-1), amino-terminal propeptide of type III procollagen (PIIINP) and hyaluronic acid (HA)
ALP response rates | Change from baseline through Week 15
  ALP response rates, defined as reduction of ALP to 1.3 x upper limit of normal (ULN), or a combination of ALP reduction to 1.5-1.3 x ULN with an at least 40%
Percent change in liver enzymes levels | Percent change from baseline through Week 15
  Percent change in liver enzymes (alanine aminotransferase [ALT]), aspartate aminotransferase [AST], and gamma glutamyl transferase [GGT])
Change in liver fibrosis markers | Change from baseline through Week 15
  Liver fibrosis markers as measured by pro-peptide of type collagen (PRO-C3) and pro-peptide of type V collagen (PRO-C5)
Elucidation of the serum Pharmacokinetics (PK) Profile - C0 | Up to 60 weeks
  Pre-dose plasma concentration
Elucidation of the serum Pharmacokinetics (PK) Profile - Cmax | Up to 60 weeks
  Observed maximum plasma concentration
Elucidation of the serum Pharmacokinetics (PK) Profile - Tmax | Up to 60 weeks
  Time to reach the observed maximum plasma concentration (Tmax)
Elucidation of the serum Pharmacokinetics (PK) Profile - AUClast | Up to 60 weeks
  Area under the plasma concentration-time curve from time of administration up to the last time point with a measurable concentration post dosing, calculated by linear up-logarithmic down trapezoidal summation.
Elucidation of the serum Pharmacokinetics (PK) Profile - AUC∞ | Up to 60 weeks
  Area under the plasma concentration-time curve extrapolated to infinity, calculated as: AUC∞ = AUClast + Clast/λz, where AUClast is the last measurable concentration.
Elucidation of the serum Pharmacokinetics (PK) Profile - λz | Up to 60 weeks
  Elimination rate constant, determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve
Elucidation of the serum Pharmacokinetics (PK) Profile - t½ | Up to 60 weeks
  Terminal elimination half-life, defined as 0.693/λz
Development of Anti-drug antibodies (ADAs) | 15 weeks
  Evaluation of the development of ADAs following repeated administration of anti-human CCL24 monoclonal antibody (CM-101)
Development of Anti-drug antibodies (ADAs) | 48 weeks
  Evaluation of the development of ADAs following repeated administration of anti-human CCL24 monoclonal antibody (CM-101)
Assessment of Pharmacodynamic (PD) parameters - Serum CCL24 levels | Up to 60 weeks
  Serum CCL24 levels
Assessment of Pharmacodynamic (PD) parameters - Inflammatory marker levels of cytokines | Up to 60 weeks
  Inflammatory marker levels of cytokines
Assessment of Pharmacodynamic (PD) parameters - Inflammatory marker levels of interleukins | Up to 60 weeks
  Inflammatory marker levels of interleukins
Assessment of Pharmacodynamic (PD) parameters - Single cell ribonucleic acid sequencing from whole blood samples | Up to 60 weeks
  Single cell ribonucleic acid sequencing from whole blood samples
Assessment of Pharmacodynamic (PD) parameters - IgG4 levels | Up to 60 weeks
  IgG4 levels will be evaluated pre-dose
Assessment of Pharmacodynamic (PD) parameters - IgG1 levels | Up to 60 weeks
  IgG1 levels will be evaluated pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frankel, MD, Study Director — ChemomAb Ltd.
Locations (33):
- United States (8):
  - Scripps Clinic Torrey Pines - site P83, La Jolla, California
  - UC Davis Health System - Midtown Ambulatory Care Center - site P79, Sacramento, California
  - Northwestern University - site P77, Chicago, Illinois
  - Massachusetts General Hospital - site P95, Boston, Massachusetts
  - Harvard Medical School - Beth Israel Deaconess Medical Center (BIDMC) - Liver Center - site P81, Boston, Massachusetts
  - Gastro One - GI Diagnostic and Therapeutic Endoscopy Center - 1310 Wolf Park - site P82, Germantown, Tennessee
  - Methodist Dallas Medical Center - site P72, Dallas, Texas
  - Virginia Commonwealth - site P94, Richmond, Virginia
- Germany (3):
  - Klinikum der Johann Wolfgang Goethe-Universitaet - site P42, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf (UKE) - site P47, Hamburg
  - Medizinische Hochschule Hannover (MHH) - site P41, Hanover
- Israel (10):
  - Soroka MC - site P23, Beersheba
  - Shamir Medical Center (Assaf Harofeh) - site P28, Be’er Ya‘aqov
  - Carmel - site P27, Haifa
  - Rambam MC - site P22, Haifa
  - Hadassah Ein Kereme - site P21, Jerusalem
  - Shaarei Tszedek Medical Center - site P29, Jerusalem
  - Galilee Medical Center - site P24, Nahariya
  - EMMS Holy Family Nazareth Hospital - site P26, Nazareth
  - Assuta Medical Center - site P31, Tel Aviv
  - Tel-Aviv Sourasky Medical Center - site P30, Tel Aviv
- Spain (4):
  - Hospital Clínic de Barcelona - site P67, Barcelona
  - Hospital Universitario Ramón y Cajal - site P61, Madrid
  - Hospital Universitari i Politècnic La Fe - site P64, Valencia
  - Hospital Universitario Miguel Servet - site P65, Zaragoza
- United Kingdom (8):
  - Leeds Teaching Hospitals NHS Trust - site P08, Leeds, WYK
  - University Hospitals Birmingham NHS Foundation Trust - site P05, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital - site P09, Cambridge
  - NHS Greater Glasgow and Clyde - site P03, Glasgow
  - King's College Hospital NHS Foundation Trust - site P04, London
  - The Royal Free Hospital - site P01, London
  - Oxford University Hospitals NHS Foundation Trust- site P11, Oxford
  - Plymouth Hospitals NHS Trust - Derriford Hospital - site P07, Plymouth